CLINICAL TRIAL: NCT06227286
Title: Enhanced External Counter Pulsation on Afterload Mismatch Rate in Post-TEER (PAMPER): A Multicenter, Randomized, Double-blind Controlled Study
Brief Title: Enhanced External Counter Pulsation on Afterload Mismatch Rate in Post-TEER (PAMPER)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Second Affiliated Hospital of Shantou University Medical College (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Zhongshan People's Hospital, Guangdong, China (Other); Jieyang People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-dong Zhuang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PAMPER Study
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EECP Arm (Experimental): Participants would be assigned for treating with EECP initiated with 0.030 MPa, 30-45 minutes per day, 5 days per week, 7 weeks in total.
  Interventions: Device: EECP
- Sham-EECP Arm (Sham Comparator): Participants would be assigned for treating with Sham-EECP initiated with 70 mmHg, 30-45 minutes per day, 5 days per week, 7 weeks in total.
  Interventions: Device: Sham-EECP

INTERVENTIONS:
Device: EECP — EECP: 30-45 minutes/day, 5 days/week, 7 weeks, initiates with 0.030MPa.
  Arms: EECP Arm
Device: Sham-EECP — EECP: 30-45 minutes/day, 5 days/week, 7 weeks, constant to 75 mmHg.
  Arms: Sham-EECP Arm

SUMMARY:
The goal of this multicenter, randomized, double-blind controlled study is to learn about the individuals after transcatheter edge-to-edge mitral valve repair (TEER). The main questions it aims to answer are: (1) can enhanced external counterpulsation (EECP) reduce the prevalence of afterload mismatch after TEER? (2) can EECP prevent the major adverse cardiac events after TEER? Participants will be randomly assigned into EECP or Sham-EECP intervention after TEER. Researchers will compare the EECP and Sham-EECP to see if it helps reduce the prevalence of afterload mismatch after TEER.

ELIGIBILITY:
Inclusion Criteria

* Consent to participate
* Age > 18 years
* Moderate or severe Mitral Regurgitation
* Patients who meet the indications for transcatheter Mitral valve edge-to-edge repair and have undergone TEERM

Exclusion Criteria

* Lower extremity deep vein thrombosis, active thrombophlebitis
* Moderate or severe aortic stenosis/insufficiency
* Moderate pulmonary hypertension (mean pulmonary pressure >50mmHg)
* Aortic aneurysm/cerebral aneurysm Uncontrolled hypertension (>180/110mmHg) Arrhythmias that may interfere with the ECG gating function of the EECP device Hemorrhagic disease or obvious bleeding tendency Limb infection Pregnant/lactating women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Afterload mismatch | Within 1 years after transcatheter Mitral valve edge-to-edge repair
  postoperative-LVEF / preoperative-LVEF <85% OR postoperative-LVEDVi / preoperative-LVEDVi >110%

SECONDARY OUTCOMES:
Major adverse composite events | Within 1 years after transcatheter Mitral valve edge-to-edge repair
  Cardiovascular death, acute heart failure, hospitalization caused by chronic heart failure, myocardial infarction, unplanned coronary revascularization (PCI/PTCA/CABGs), stroke

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Zhuang, PhD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (6):
- China (6):
  - First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Third Affiliated Hospital, Sun Yat-Sun University, Guangzhou, Guangdong
  - Jieyang People's Hospital, Jieyang, Guangdong
  - Second Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong